CLINICAL TRIAL: NCT07289945
Title: A COMPARATIVE STUDY OF DESFLURANE VERSUS SEVOFLURANE IN ELDERLY PATIENTS: EFFECT ON EARLY RECOVERY
Brief Title: Effects of Sevoflurane vs Desflurane on Early Recovery and Cognitive Function in Elderly Patients Undergoing Scheduled Non-Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, jebri alia, Head of Anesthesiology and Intensive Care Department at Charles Nicolle Hospital in Tunis, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWA 00032748 IORG0011243
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Early Recovery in Elderly Patients; Cognitive Function
Keywords: desflurane; sevoflurane; elderly; general anesthesia; recovery; cognition
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Intervention Model Description: This prospective randomized single-blind trial compares desflurane versus sevoflurane for assessing early postoperative recovery and cognitive function in elderly patients undergoing elective non-cardiac surgery. Primary objectives: evaluate the time from discontinuation of the volatile agent to eye opening, response to verbal commands, and extubation. Secondary objectives include the time required to achieve a modified Aldrete Score (MAS) ≥9, post-anesthesia care unit (PACU) discharge time, and the interval to reach an SOMCT score ≥20. Inclusion criteria: patients aged over 60 years, ASA physical status I-III, scheduled for elective non-cardiac surgery under general anesthesia. Exclusion criteria: pre-existing cognitive impairment (baseline SOMCT <20), severe hepatic or renal failure, anticipated difficult airway, emergency surgery, or refusal to participate. A total of 81 patients were randomized into two groups to receive either desflurane or sevoflurane for anesthesia maintenance.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane group (Active Comparator): Participants receive Sevoflurane for anesthesia maintenance with a Fresh Gaz Flow of less than 1 L/min.
  Interventions: Drug: Sevoflurane
- Desflurane group (Active Comparator): Participants receive Desflurane for anesthesia maintenance with a Fresh Gaz Flow of less than 0.5 L/min.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane used for anesthesia maintenance with a MAC of 2-3% and FGF of less than 1 L/min.
  Arms: sevoflurane group
Drug: Desflurane — Desflurane used for anesthesia maintenance with a MAC of 4-6% and FGF of less than 0.5 L/min.
  Arms: Desflurane group

SUMMARY:
The goal of this clinical study is to compare the effects of desflurane versus sevoflurane on early postoperative recovery and cognitive function in elderly patients (aged 60 years and older, ASA I-III) undergoing elective non-cardiac surgery under general anesthesia. The main questions this study aims to answer are:

Which anesthetic agent allows faster emergence from anesthesia (eye opening, response to commands, extubation)? Does desflurane lead to earlier cognitive recovery as measured by the Short Orientation Memory Concentration Test (SOMCT)? Does the choice of volatile anesthetic influence the time required to achieve a modified Aldrete score (MAS) ≥ 9 and PACU discharge readiness? Researchers compared the desflurane group to the sevoflurane group to determine whether desflurane provides a superior recovery profile and minimizes delayed emergence in elderly surgical patients.

Participants will:

Be randomly assigned to receive either desflurane or sevoflurane for maintenance of general anesthesia.

Undergo standardized induction with fentanyl, propofol, and cisatracurium, along with uniform ventilatory and monitoring protocols.

Have emergence parameters recorded immediately after discontinuation of the inhaled agent (eye opening, command following, extubation).

Be evaluated in the post-anesthesia care unit using the modified Aldrete Score (MAS) and SOMCT, with predefined thresholds for recovery (MAS ≥ 9, SOMCT ≥ 20). This study aims to determine whether desflurane-due to its lower blood/gas partition coefficient-offers measurable clinical benefits in terms of rapid awakening, cognitive recovery, and overall early postoperative recovery in the geriatric population.

DETAILED DESCRIPTION:
Delayed emergence from anesthesia and early postoperative cognitive decline represent important clinical challenges in elderly surgical patients, who commonly exhibit reduced physiological reserve, altered pharmacodynamics, and multiple comorbidities. The combination of age-related organ changes, diminished drug clearance, and increased sensitivity of the central nervous system places this population at heightened risk of prolonged awakening, impaired reflexes, and postoperative disorientation. Volatile anesthetics such as sevoflurane and desflurane are widely used in geriatric anesthesia owing to their low blood/gas solubility and generally favorable recovery profiles, yet their comparative impact on early emergence and cognitive recovery remains insufficiently established. This prospective randomized single-blind trial is therefore designed to compare desflurane with sevoflurane in elderly patients undergoing elective non-cardiac surgery, with the objective of determining whether desflurane's lower blood/gas partition coefficient translates into clinically meaningful improvements in postoperative recovery.

Conditions Conditions: Postoperative Delayed Emergence and Early Cognitive Decline in Elderly Surgical Patients Keywords: general anesthesia, elderly, desflurane; sevoflurane; recovery, cognition. Study Design Study Type: Interventional. The perioperative protocol begins with standard patient preparation, including verification of the pre-anesthesia checklist and initiation of monitoring with ECG, pulse oximetry, non-invasive blood pressure, and capnography. Three baseline hemodynamic readings are recorded to establish reference values. Two peripheral IV lines (18-20G) are inserted for fluids and medication administration. Patients underwent a baseline Short Orientation Memory Concentration Test (SOMCT). Anesthesia induction is standardized with Fentanyl: 2 µg/kg, Propofol: titrated to loss of consciousness, Cisatracurium: 0.15 mg/kg to facilitate intubation. Endotracheal intubation is confirmed by capnography. Patients are randomized into two groups:

Group D - Desflurane, Group S - Sevoflurane, maintenance protocol under controlled ventilation targeting ETCO₂ between 30 and 40 mmHg. Volatile agents are discontinued at the end of surgery, and emergence parameters-including time to eye opening, response to verbal commands, and extubation-were recorded by a blinded observer. In the post-anesthesia care unit, recovery is assessed using the modified Aldrete Score (MAS) until ≥9 and SOMCT until ≥20, and discharge times are documented. Hemodynamic, respiratory, and anesthetic variables are continuously monitored throughout the procedure. Statistical Analysis: Data entry and analysis will be performed using SPSS software (version 25.0). Descriptive Analysis: Normally distributed continuous quantitative variables will be summarized as mean ± standard deviation. Non-normally distributed continuous variables will be reported as median and interquartile range [IQR: 25%-75%]. Categorical variables will be presented as absolute frequencies (n) and relative frequencies (%). Analytical Analysis: Associations between two categorical variables will be assessed using Pearson's chi-square test when conditions are met; otherwise, Fisher's exact test will be applied. For comparisons between a categorical and a normally distributed quantitative variable, Student's t-test will be used, while the Mann-Whitney U test will be employed for non-parametric data. A significance level of p < 0.05 will be considered statistically significant. In multivariate analysis, risk estimates will be expressed as odds ratios (OR) with 95% confidence intervals (95% CI).

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients whose ages are superior to 60 years of age [1].
* Patients with an American Society of Anesthesiologists Classification (ASA) I, II or III stable (Annex 1).
* Patients undergoing elective non-cardiac surgery under general anesthesia with tracheal intubation.

Non-inclusion criteria:

* Patients having declined to participate in the study protocol.
* Patients with a contraindication for minimal flow anesthesia such as hyperthermia, smoke intoxication and ketoacidosis metabolic condition (for example, anorexia nervosa).
* Patients with history of malignant hyperthermia.
* Patients with Psychotic disorders.
* Patients with substance abuse.
* Patients with severe obstructive or restrictive pulmonary disease.
* Patients with hepatic disease.
* Patients with end stage renal disease.
* Patients with history of allergy to study drugs.

Exclusion Criteria:

* We excluded from our study patients who presented with perioperative complication or instability requiring ICU transfer due to extubation failure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Time to eye opening | within 3 to 24 minutes after discontinuiation of the volatile agent
  Time from discontinuation to the volatile agent to eye opening
Time to obey verbal command | within 5 to 40 minutes after discontinuation of the volatile agent
  Time from discontinuation of the volatile agent to obeying verbal command
Time to extubation | within 6 to 30 minutes after disontinuation of the volatile agent
  Time from discontinuation of the volatile agent to extubation

SECONDARY OUTCOMES:
Time to reach a Modified Aldrete Score 9 or greater | within 10 to 48 minutes after discontinuation of the volatile agent
  Time from discontinuation of the volatile agent to reaching a Modified Aldrete Score 9 or greater
Time to discharge from the recovery room | within 12 to 53 minutes after discontinuation of the volatile agent
  Time from discontinuation of the volatile agent to discharge from the recovery room
Time to reach a SOMCT 20 or higher | within 15 to 55 minutes from discontinuation of the volatile agent
  Time from discontinuation of the volatile agent to reaching a SOMCT 20 or higher

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Charles Nicolle, Tunis, Tunis 1006, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim CT, Myung W, Lewis M, Lee H, Kim SE, Lee K, Lee C, Choi J, Kim H, Carroll BJ, Kim DK. Exposure to General Anesthesia and Risk of Dementia: A Nationwide Population-Based Cohort Study. J Alzheimers Dis. 2018;63(1):395-405. doi: 10.3233/JAD-170951. PMID 29614656
- [Background] Katzman R, Brown T, Fuld P, Peck A, Schechter R, Schimmel H. Validation of a short Orientation-Memory-Concentration Test of cognitive impairment. Am J Psychiatry. 1983 Jun;140(6):734-9. doi: 10.1176/ajp.140.6.734. PMID 6846631
- [Background] Jindal R, Kumra VP, Narani KK, Sood J. Comparison of maintenance and emergence characteristics after desflurane or sevoflurane in outpatient anaesthesia. Indian J Anaesth. 2011 Jan;55(1):36-42. doi: 10.4103/0019-5049.76604. PMID 21431051
- [Background] Kaur A, Jain AK, Sehgal R, Sood J. Hemodynamics and early recovery characteristics of desflurane versus sevoflurane in bariatric surgery. J Anaesthesiol Clin Pharmacol. 2013 Jan;29(1):36-40. doi: 10.4103/0970-9185.105792. PMID 23493107
- [Background] Saha M, Saxena KN, Wadhwa B. Comparative study of recovery of airway reflexes and cognitive function following sevoflurane versus desflurane anaesthesia. Indian J Anaesth. 2021 Apr;65(4):282-288. doi: 10.4103/ija.IJA_1219_20. Epub 2021 Apr 15. PMID 34103741
- [Background] La Colla L, Albertin A, La Colla G, Mangano A. Faster wash-out and recovery for desflurane vs sevoflurane in morbidly obese patients when no premedication is used. Br J Anaesth. 2007 Sep;99(3):353-8. doi: 10.1093/bja/aem197. Epub 2007 Jul 9. PMID 17621601
- [Background] White PF, Tang J, Wender RH, Yumul R, Stokes OJ, Sloninsky A, Naruse R, Kariger R, Norel E, Mandel S, Webb T, Zaentz A. Desflurane versus sevoflurane for maintenance of outpatient anesthesia: the effect on early versus late recovery and perioperative coughing. Anesth Analg. 2009 Aug;109(2):387-93. doi: 10.1213/ane.0b013e3181adc21a. PMID 19608808
- [Background] Gangakhedkar GR, Monteiro JN. A prospective randomized double-blind study to compare the early recovery profiles of desflurane and sevoflurane in patients undergoing laparoscopic cholecystectomy. J Anaesthesiol Clin Pharmacol. 2019 Jan-Mar;35(1):53-57. doi: 10.4103/joacp.JOACP_375_17. PMID 31057241
- [Background] Wang C, Li L, Xu H, Lv H, Zhang H. Effect of desflurane-remifentanil or sevoflurane-remifentanil on early recovery in elderly patients: a meta-analysis of randomized controlled trials. Pharmazie. 2019 Apr 1;74(4):201-205. doi: 10.1691/ph.2019.8935. PMID 30940302
- [Background] Lockwood G. Theoretical context-sensitive elimination times for inhalation anaesthetics. Br J Anaesth. 2010 May;104(5):648-55. doi: 10.1093/bja/aeq051. Epub 2010 Mar 16. PMID 20233751
- [Background] Wagner S, Breitkopf M, Ahrens E, Ma H, Kuester O, Thomas C, von Arnim CAF, Walther A. Cognitive function in older patients and their stress challenge using different anesthesia regimes: a single center observational study. BMC Anesthesiol. 2023 Jan 6;23(1):6. doi: 10.1186/s12871-022-01960-7. PMID 36609226
- See also: World Health Organization. World Health Statistics 2016: Monitoring Health for the Sustainable Development Goals — https://www.who.int/publications/i/item/9789241565264
- See also: National Library of Medicine. Sevoflurane [Online]. Bethesda (MD): National Center for Biotechnology Information — https://pubchem.ncbi.nlm.nih.gov/compound/5206
- See also: Effect of desflurane and sevoflurane on postoperative cognitive dysfunction: A meta-analysis of randomized controlled trials — https://assets-eu.researchsquare.com/files/rs-2655326/v1/c05e153e-64fa-4db4-8fbe-6b8d8b5ed052.pdf?c=1681836278